CLINICAL TRIAL: NCT05201482
Title: Assessing the Impact of a Head-mounted Augmented Reality Low Vision Aid on Vision and Quality of Life in Children and Young People With Visual Impairment
Brief Title: Assessment of an Augmented Reality Low Visual Aid in Children and Young People With Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH-2551
Record Dates: First submitted 2021-06-04; First posted 2022-01-21 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Vision Disability
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 25 patients aged 8-16 years with moderate or severe visual impairment (Experimental): 25 patients aged 8-16 years with moderate or severe visual impairment will test the impact of a head-mounted augmented reality low vision aid (SightPlus) on vision and quality of life
  Interventions: Device: SightPlus

INTERVENTIONS:
Device: SightPlus — SightPlus is a head-mounted, augmented reality low vision aid. SightPlus enables people with a visual impairment to use their remaining vision to see more clearly up close and at a distance. SightPlus is commercially available, non-invasive, CE marked, and a MHRA approved class 1 medical device.

SUMMARY:
Approximately 24,500 children and young people (CYP) in England have a visual impairment (VI). VI refers to a loss of vision that cannot be corrected with glasses or contact lenses.

Low vision aids (e.g. magnifying glasses) can help CYP with a VI see more clearly. However, current low vision aids are not suitable for many of the activities CYP regularly engage in, such as watching TV or school lessons.

SightPlus is an advanced head-mounted digital low vision aid for CYP and adults. SightPlus helps people with a VI use their remaining vision to see more clearly up close and at a distance.

SightPlus was recently tested at Moorfields Eye Hospital in London with 60 adults with a VI. The results showed that adults could see more clearly while using SightPlus.

The study proposed here aims to find out whether SightPlus can improve the vision and quality of life of CYP aged 8-16 years with a VI.

For this study, 25 CYP will come to Sheffield Children's Hospital (SCH) for an 80-minute session with parents/guardians where they will have their vision tested, complete questionnaires measuring their vision-related quality of life and functional vision (i.e. what someone can see), and learn how to use SightPlus.

CYP will then be asked to use SightPlus for four weeks. Parents/guardians will record the activities CYP use SightPlus for in a home diary.

After four weeks, CYP and their parents/guardians will come back to SCH for a 90-minute session where they will have their vision tested with and without SightPlus, complete another vision-related quality of life and functional vision questionnaire, hand in their home diary, and complete a feedback form about their experiences of using SightPlus.

This study will help us find out whether SightPlus can improve the vision and quality of life of CYP with a VI.

DETAILED DESCRIPTION:
This study aims to assess the impact of a head-mounted augmented reality low vision aid (SightPlus) on vision and quality of life in CYP aged 8-16 years with moderate or severe VI.

There are 24,500 children and young people (CYP) with a moderate or severe visual impairment (VI) in England, of which 9,535 are registered as blind or partially sighted. CYP with VI have to live with sight loss that significantly impacts their daily lives. VI often has adverse effects on CYP's social, educational, psychological, and physical development and quality of life.

CYP with a moderate or severe VI have some vision but the image can be very blurry. Low vision aids (e.g. optical magnifiers) can improve CYP's functional vision (i.e. what an individual can actually see). Low vision aids therefore have the potential to significantly improve independent living, access to education/work, and quality of life.

However, current low vision aids are very limited in their functionality. For instance, optical magnifiers require the user to place the device over a section of text and bend over to read the magnified text. Current low vision aids are therefore largely unsuitable for the types of activities CYP typically engage in, such as school lessons, playing a musical instrument, and socialising with friends and family. There is a clear need for innovative low vision aids for CYP with VI.

SightPlus is a hands-free, head-mounted, digital low vision aid for CYP and adults with VI. SightPlus combines augmented and virtual reality by using the backlit screen of a mobile phone, placed inside a virtual reality headset, to display augmented imagery of what the user is looking at. SightPlus has various modes depending on the user's needs and enables users to see clearly both up close and at a distance. Thus, SightPlus enables individuals to use their residual sight to regain functional vision, empowering users to engage in a wide range of daily activities.

In 2017, GiveVision conducted a pilot study to assess the functionality, usability, and acceptability of SightPlus. 194 individuals (including 23 CYP aged 8-16 years) participated in a 1:1 training session. Following this session, participants were given the opportunity to trial the device at home for 2 weeks. 87% of CYP (20/23) participated in the two-week trial. During the trial, 75% of CYP used SightPlus for schoolwork and reported that school was a deciding factor in wanting to keep the device. 70% of CYP also used SightPlus for hobbies, including watching TV, playing games, reading, and playing a musical instrument. Critically, 6-9 months later, 71% of CYP still used SightPlus daily and 80% reported having greater independence and being able to do activities they were previously unable to do (e.g. reading normal print books).

GiveVision subsequently conducted a clinical study in collaboration with Moorfields Eye Hospital NHS Foundation Trust. This study examined the impact of SightPlus on visual acuity (i.e. clarity of vision) and contrast sensitivity (i.e. ability to distinguish an object from its background) in 60 adults with moderate or severe VI. After a one-hour training session, SightPlus was found to significantly improve visual acuity and contrast sensitivity, and participants reported that they would like to use the device for watching TV, reading, education, and going to the theatre/cinema.

The study proposed here aims to build on and extend the work conducted so far to assess whether a head-mounted augmented reality low vision aid can clinically improve vision and vision-related quality of life in CYP with moderate or severe VI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-16 years
* Corrected visual acuity equal to lower than 6/18 and equal to or better than 3/60 with both eyes open
* Central vision loss or vision loss affecting the whole visual field
* Currently cared for by the Eye Department at Sheffield Children's Hospital
* Patient and parents/guardians fluent in verbal and written English
* No physical or cognitive difficulties which indicate the child or young person would struggle to use device or complete the study activities

Exclusion Criteria:

* Aged <8 years or >17 years
* Corrected visual acuity not lower than 6/18 or equal to or better than 3/60 with both eyes open
* History of neurological conditions, such as epilepsy or seizures
* Children with a pacemaker or other implanted medical device
* Not currently cared for by the Eye Department at Sheffield Children's Hospital
* Patients or parents/guardian non-fluent in verbal and written English
* Physical or cognitive difficulties which indicate the child or young person would struggle to use device or complete the study activities

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Assess change in maximum reading speed in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Maximum reading speed will be assessed using MNRead
Assess change in reading acuity in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Reading acuity will be assessed using MNRead
Assess change in binocular visual acuity in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Binocular visual acuity will be measured using Keeler Crowded logMAR
Assess change in near visual acuity in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Near visual acuity will be measured using Sloan reduced logMAR
Assess change in contrast sensitivity in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Contrast Sensitivity will be measured using the Evans Low Contrast Sensitivity test
Assess change in facial expressions in patients aged 8-16 years with moderate or severe visual impairment | Perform test at first study visit (50 min duration), then let the patient use the SightPlus device for four weeks and then perform test again at the second study visit (70 min duration)
  Facial expressions will be assessed using the NimStim Dataset and the number of errors will be counted
Assess change in vision-related quality of life in patients aged 8-16 years with moderate or severe visual impairment | Ask patients to complete the baseline questionnaire immediately after the first visit at home and to complete the post-trial questionnaire at home at end of the four week trial period (with the Sightplus device) and return this at the 2nd clinic visit
  Patients will asked to complete baseline and post-trial vision-related quality of life questionnaires.
Assess change in functional vision in patients aged 8-16 years with moderate or severe visual impairment | Ask patients to complete the baseline questionnaire immediately after the first visit at home and to complete the post-trial questionnaire at home at end of the four week Sightplus device trial period and return this at the 2nd clinic visit
  Patients will asked to complete baseline and post-trial functional vision questionnaires.
Determine how and when patients aged 8-16 years with moderate or severe visual impairment use the SightPlus device | The home diary is completed by the patient at home during the four week trial of the SightPlus device when it is used. The home diary is returned during the second visit to the clinic
  Patients will be given a home diary to complete during the four week trial using the SightPlus device.
Determine usability and acceptability of Sightplus device | Patients and parents/carers will be given usability/acceptability feedback form to complete at home at the end of the four-week trial period. They will return this at the second clinic visit
  Patients and parents/carers will be given a usability/acceptability feedback form to complete

CONTACTS AND LOCATIONS:
Overall Officials: Finnguala Burgum, Principal Investigator — Sheffield Children's NHS Foundation Trust
Locations (1):
- Clinical Research Facility, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: No